CLINICAL TRIAL: NCT03058081
Title: Acute Effects of High Flow Nasal Support During Exercise in Patients With COPD After Severe Exacerbation
Brief Title: Effect of High Flow Nasal During Exercise in COPD Patients
Acronym: AiRehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01325-46
Record Dates: First submitted 2017-01-23; First posted 2017-02-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: COPD Exacerbation
Keywords: COPD; Exercise; High Flow Nasal; Muscle Oxygenation; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Test (Experimental): Patients will perform one Constant Work-Rate Exercise Test at 80% of maximum workload with High Flow Nasal at 60L/min (with or without additional oxygen)
  Interventions: Device: High Flow nasal cannula
- Control Test (No Intervention): Patient will perform one Constant Work-Rate Exercise Test at 80% of maximum workload on room air or with oxygen supplementation

INTERVENTIONS:
Device: High Flow nasal cannula — High intensity Constant Work-Rate exercise test with High Flow Nasal Cannula in COPD patients involved in a Pulmonary Rehabilitation Program after an exacerbation (< 7 days after hospital discharge). High Flow nasal will be administered through nasal cannula using the Airvo2 (Fisher&Paykel)
  Arms: High Flow Nasal Test

SUMMARY:
Early pulmonary rehabilitation is recommended after an episode of severe exacerbation of chronic obstructive pulmonary disease (COPD). However, its implementation is challenging particularly as regard exercise training. High flow ventilation in reducing work of breathing and dyspnea may improve exercise tolerance. The aim of this study is to carry out the acute effect of high flow nasal cannula on exercise endurance in post-exacerbation copd patients

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of COPD

Exclusion Criteria:

* exercise contraindication Any musculoskeletal problems, cardiovascular or neurological comorbidities that limits exercise.
* pH < 7,35
* Body temperature > 38°C
* cardiac frequency > 100 bpm at rest
* systolic blood pressure < 100 mmHg
* exacerbation during the study

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Difference in exercise capacity | The outcome will be measure after every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 3 days maximum
  Difference in endurance time (TLim) during High Intensity Constant Work-Rate Endurence Test (CWRET)

SECONDARY OUTCOMES:
Difference in peripheral muscle oxygenation | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 3 days maximum. Data will be continuously collected during exercise
  Muscle oxygenation will be evaluated using Near-infrared spectroscopy technology.
Difference in Dyspnea and muscular fatigue | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 3 days maximum. Data will be collected every 2 minute during tests and at the end of the exercise
  Difference in dyspnea and muscular fatigue using Modified Borg Scale (0 - 10 points)
Difference in Oxygen Saturation | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 3 days maximum. Data will be continuously collected during exercise
  Difference in Oxygen Saturation using a pulse oximetry (SpO2)
Difference in Cardiac Frequency | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 3 days maximum. Data will be continuously collected during exercise
  Difference in Cardiac Frequence using a pulse oximetry
Difference in Transcutaneous Carbon Dioxide | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 3 days maximum. Data will be continuously collected during exercise
  Difference Transcutaneous Carbon Dioxide using Transcutaneous Carbon Dioxide using a Transcutaneous capnography
Difference in Respiratory Rate | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 3 days maximum. Data will be continuously collected during exercise
  Difference in Respiratory Rate using a Respiratory Inductive Plethysmography
Difference in Respiratory Muscle Fatigue | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 3 days maximum. Data will be collected before and 5 minute maximum after exercise
  Difference in Respiratory Muscle Fatigue using an electronical manometer

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier du Havre, Montivilliers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prieur G, Medrinal C, Combret Y, Dupuis Lozeron E, Bonnevie T, Gravier FE, Quieffin J, Lamia B, Borel JC, Reychler G. Nasal high flow does not improve exercise tolerance in COPD patients recovering from acute exacerbation: A randomized crossover study. Respirology. 2019 Nov;24(11):1088-1094. doi: 10.1111/resp.13664. Epub 2019 Aug 6. PMID 31387158
- [Derived] Prieur G, Medrinal C, Combret Y, Quesada AR, Prieur F, Quieffin J, Borel JC, Reychler G. Effect of high-flow nasal therapy during acute aerobic exercise in patients with chronic obstructive pulmonary disease after exacerbation: protocol for a randomised, controlled, cross-over trial. BMJ Open Respir Res. 2017 Aug 16;4(1):e000191. doi: 10.1136/bmjresp-2017-000191. eCollection 2017. PMID 29071072